CLINICAL TRIAL: NCT03315559
Title: An Open-label Study in Healthy Male Subjects, to Determine the Excretion Balance and Pharmacokinetics of [14C]-GSK2269557, Administered as a Single Intravenous Microtracer (Concomitant With an Inhaled Non-radiolabelled Dose) and a Single Oral Dose
Brief Title: Absorption & Elimination of Radiolabelled GSK2269557
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 206764; 2017-002347-16 (EudraCT Number)
Record Dates: First submitted 2017-10-17; First posted 2017-10-20 (Actual); Results first posted 2019-03-20 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: GSK2269557; Pharmacokinetics; Radiolabel; Healthy; Excretion; Bioavailability
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: This will be a 2-period, single-sequence crossover study. Subjects will receive IV and inhaled doses of GSK2269557 in treatment period 1 and oral dose of GSK2269557 in treatment period 2.
Masking Description: This will be an open-label study. Hence, masking will not be provided to the subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subjects receiving GSK2269557 in treatment period 1 (Experimental): Eligible subjects will receive IV infusion of [14C] radiolabelled GSK2269557 with a single dose of 10 micrograms (µg) administered as single microtracer, concomitantly with an inhaled nonradiolabelled 1000 µg dose of GSK2269557. There will be a washout of at least 14 days after inhaled and IV dosing before subjects receive treatment 2.
  Interventions: Drug: [14C]-GSK2269557 IV infusion; Drug: GSK2269557 via DPI; Drug: [14C]-GSK2269557 oral solution
- Subjects receiving GSK2269557 in treatment period 2 (Experimental): Eligible subjects will receive [14C]-GSK2269557 with a single dose of 800 µg, administered as an oral solution.
  Interventions: Drug: [14C]-GSK2269557 IV infusion; Drug: GSK2269557 via DPI; Drug: [14C]-GSK2269557 oral solution

INTERVENTIONS:
Drug: [14C]-GSK2269557 IV infusion — The [14C]-GSK2269557 solution will be available in dosing strength of 10 µg, administered as single dose IV infusion over 15 minutes. It will be prepared by dissolving a hemisuccinate salt (GSK2269557T) in normal saline.
Drug: GSK2269557 via DPI — GSK2269557 DPI will be available with dosing strength of 1000 µg, administered as oral inhalation intended to inhale twice. It will be prepared by blending GSK2269557 hemisuccinate salt (GSK2269557H) with lactose and magnesium stearate.
Drug: [14C]-GSK2269557 oral solution — The [14C]-GSK2269557 solution will be available with dosing strength of 800 µg, administered as single dose orally. It will be prepared by dissolving [14C]-GSK2269557 hemisuccinate salt (GSK2269557T) in water.

SUMMARY:
GSK2269557 is being developed as an anti-inflammatory agent for the treatment of chronic obstructive pulmonary disease (COPD) and other inflammatory lung diseases such as asthma. This study is designed to investigate the recovery, excretion, and pharmacokinetics (PK) of (14 Carbon [C])-GSK2269557 administered as a single intravenous (IV) dose (concomitant with an inhaled non-radiolabelled dose) and as a single oral dose in 6 healthy male subjects. Subjects will receive [14C] radiolabelled GSK2269557 administered as IV infusion, with a nonradiolabelled dose of GSK2269557 via dry powder inhaler (DPI) in treatment period 1 and a single dose of [14C]-GSK2269557, administered as an oral solution in treatment period 2. There will be a washout period of at least 14 days after inhaled and IV dosing before subjects takes part in treatment period 2. The IV microtracer dose of GSK2269557 will be administered concomitant to an inhaled non-radiolabelled dose to ensure that the pharmacokinetics represent a clinically relevant dose. The total study duration will be up to 11 weeks, including a screening visit, 2 treatment periods and a follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 30 to 55 years of age inclusive, at the time of signing the informed consent.
* Subjects who are overtly healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, vital signs, laboratory tests, and cardiac monitoring; A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator agrees and documents that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* A history of regular bowel movements (averaging one or more bowel movements per day).
* Body weight >= 50 kilograms (Kg) and body mass index (BMI) within the range 19.0-31.0 kg per meter square (kg/m^2) (inclusive).
* Male subjects will be included.
* Subjects with female partners of childbearing potential must agree to use contraception during the treatment period, from the time of first dose of study medication until follow-up, and refrain from donating sperm during this period.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Alanine aminotransferase (ALT) > 1.5x Upper limit of normal (ULN).
* Bilirubin > 1.5xULN (isolated bilirubin > 1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Mean QT duration corrected for heart rate by Fridericia's formula (QTCF) > 450 milliseconds (msec).
* Any clinically relevant abnormality identified at the screening medical assessment (physical examination/medical history), clinical laboratory tests, or 12-lead ECG.
* A pre-existing condition(s) interfering with normal gastrointestinal (GI) anatomy or motility, including constipation, malabsorption or other GI dysfunction which may interfere with the absorption, distribution, metabolism or elimination of the study drug. Subjects with a history of cholecystectomy must be excluded.
* At screening, a supine or semi-supine BP that is persistently higher (triplicate measurements at least 2 minutes apart than 140/90 millimeters of mercury (mmHg).
* At screening, a supine or semi-supine mean heart rate (HR) outside the range 40-90 beats per minute (BPM).
* Subject is mentally or legally incapacitated.
* A history of respiratory disease (example given [e.g.] history of asthma) in the last 10 years.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) before the first dose of study medication, unless in the opinion of the investigator and GlaxoSmithKline (GSK) Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* Need of Paracetamol or Acetaminophen, at doses of > 2 grams (g)/day. Other concomitant medication may be considered on a case by case basis by the GSK Medical Monitor.
* The subject has participated in a clinical trial and has received an investigational product (IP) within 3 months before their first dose in the current study.
* Participation in a clinical trial involving administration of 14C-labelled compound(s) within the last 12 months. A subject's previous effective dose will be reviewed by the medical investigator to ensure there is no risk of contamination/carryover into the current study.
* Presence of hepatitis B surface antigen (HBsAg), or positive hepatitis C antibody test result at screening.
* Positive Hepatitis C ribonucleic acid (RNA) test result at screening or within 3 months prior to first dose of study treatment.
* A positive test for Human Immunodeficiency Virus (HIV) antibody.
* A positive pre-study drug/alcohol screen.
* Exposure to more than four new chemical entities within 12 months before the subject's first dose.
* Subjects have received a total body radiation dose of greater than 5.0 micro sievert (mSv) (upper limit of World Health Organization [WHO] category II) or exposure to significant radiation (e.g. serial x-ray or computed tomography [CT] scans, barium meal etc) in the 12 months before this study.
* An occupation which requires monitoring for radiation exposure, nuclear medicine procedures or excessive x-rays within the past 12 months.
* Participation in the study would result in donation of blood or blood products in excess of 500 milliliters (mL) within a 90 day period.
* Unwillingness or known inability to follow the procedures outlined in the protocol, including the use of the Enterotest capsule.
* History of regular alcohol consumption within 6 months of the study, defined as an average weekly intake of >21 units. One unit is equivalent to 8 g of alcohol: a halfpint (approximately 240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Urinary cotinine levels indicative of smoking; current smoker; or ex-smokers who gave up less than 6 months ago or who have a history of more than 10 pack-years. Pack-years = cigarettes per day x number of years smoked/20

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study will include 6 healthy male subjects.
Enrollment: 6 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2017-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20278

REFERENCES:
- [Background] Harrell AW, Wilson R, Man YL, Riddell K, Jarvis E, Young G, Chambers R, Crossman L, Georgiou A, Pereira A, Kenworthy D, Beaumont C, Marotti M, Wilkes D, Hessel EM, Fahy WA. An Innovative Approach to Characterize Clinical ADME and Pharmacokinetics of the Inhaled Drug Nemiralisib Using an Intravenous Microtracer Combined with an Inhaled Dose and an Oral Radiolabel Dose in Healthy Male Subjects. Drug Metab Dispos. 2019 Dec;47(12):1457-1468. doi: 10.1124/dmd.119.088344. Epub 2019 Oct 24. PMID 31649125

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at a single center in the United Kingdom from 14-November-2017 to 22-December-2017.
Pre-assignment Details: A total of 7 participants were screened, of which 1 participant was a reserve participant and was not used. The remaining 6 participants were enrolled.
Groups:
- All Study Participants: Participants received intravenous (IV) infusion of [14C] radiolabeled GSK2269557 along with a single dose of 10 micrograms (µg) administered as single microtracer, concomitantly with an inhaled non-radiolabeled 1000 µg dose of GSK2269557 in Treatment Period 1. There was a washout of at least 14 days. Participants received [14C]-GSK2269557 with a single dose of 800 µg, administered as an oral solution in Treatment Period 2.
Period: Treatment Period 1 (8 Days)
Arm/Group | All Study Participants
Started | 6
Completed | 6
Not Completed | 0
Period: Washout Period (14 Days)
Arm/Group | All Study Participants
Started | 6
Completed | 6
Not Completed | 0
Period: Treatment Period 2 (15 Days)
Arm/Group | All Study Participants
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: Years] — Safety Population comprised of all participants in the All Participants Enrolled (APE) Population (All participants for whom a record exists on the study database; included both screened and unscreened participants but signed the informed consent form) who received at least one dose of study treatment.
  Years | 43.3 (10.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Race/Ethnicity, Customized [Number; unit: Count of participants]
  African American/African Heritage | 2
  White - White/Caucasian/European Heritage | 4

OUTCOME MEASURES:

1. Primary Outcome: Area Under Concentration-time Curve (AUC) From Time 0 (Pre-dose) to Infinite Time (0 to Inf) and AUC From Time 0 (Pre-dose) to Last Time of Quantifiable Concentration (0 to t) of Total Drug-related Material (Radioactivity) in Plasma for Treatment Period 1
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis. Pharmacokinetic (PK) Population comprised of participants in the APE Population who received at least one dose of study treatment and for whom a PK sample was obtained and analyzed. Only those participants available at the specified time points were analyzed represented by n=X in the category titles.
Time Frame: Pre-dose and at 0 hour (post inhalation and pre-IV infusion), at the end of infusion and at 0.33, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96 and 168 hours after the start of infusion
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*picogram Equivalent per millilitre
Groups:
- Nemi IH + 14C-Nemi IV: Participants received IV infusion of [14C] radiolabeled GSK2269557 as a single dose of 10 µg administered as single microtracer, concomitantly with an inhaled non-radiolabeled 1000 µg dose of GSK2269557.
Arm/Group | Nemi IH + 14C-Nemi IV
Number analyzed (Participants) | 6
Hour*picogram Equivalent per millilitre
  AUC (0 to inf), n=3: number analyzed (Participants) | 3
  AUC (0 to inf), n=3 | 812.8550 (8.17885)
  AUC (0 to t), n=6 | 770.3316 (17.70272)

2. Primary Outcome: AUC From Time Zero (Pre-dose) Extrapolated to Infinite Time (0 to Inf) and AUC From Time Zero (Pre-dose) to Last Time of Quantifiable Concentration (0 to t) of Total Drug-related Material (Radioactivity) in Plasma for Treatment Period 2
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis. Only those participants available at the specified time points were analyzed represented by n=X in the category titles. NA indicates that data is not available as single participant was analyzed.
Time Frame: Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96 and 168 h post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*picogram Equivalent per millilitre
Groups:
- 14C-Nemi Oral: Participants received [14C]-GSK2269557 as a single dose of 800 µg, administered as an oral solution.
Arm/Group | 14C-Nemi Oral
Number analyzed (Participants) | 6
Hour*picogram Equivalent per millilitre
  AUC (0 to inf), n=1: number analyzed (Participants) | 1
  AUC (0 to inf), n=1 | 34749.40 (NA) — NA indicates that data is not available as single participant was analyzed
  AUC (0 to t), n=6 | 31730.13 (35.715)

3. Primary Outcome: Maximum Observed Concentration (Cmax) of Total Drug-related Material (Radioactivity) in Plasma for Treatment Period 1
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis.
Time Frame: as for outcome 1
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram Equivalent per milliliter
Arm/Group | Nemi IH + 14C-Nemi IV
Number analyzed (Participants) | 6
Picogram Equivalent per milliliter | 204.4057 (52.32698)

4. Primary Outcome: Cmax of Total Drug-related Material (Radioactivity) in Plasma for Treatment Period 2
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis.
Time Frame: Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96 and 168 h post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram Equivalent per milliliter
Arm/Group | 14C-Nemi Oral
Number analyzed (Participants) | 6
Picogram Equivalent per milliliter | 703.5192 (24.43331)

5. Primary Outcome: Time of Occurrence of Cmax (Tmax) of Total Drug-related Material (Radioactivity) in Plasma for Treatment Period 1
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis.
Time Frame: as for outcome 1
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Nemi IH + 14C-Nemi IV
Number analyzed (Participants) | 6
Hours | 0.2333 [0.2333 to 0.2333]

6. Primary Outcome: Tmax of Total Drug-related Material (Radioactivity) in Plasma for Treatment Period 2
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis.
Time Frame: Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96 and 168 h post-dose
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | 14C-Nemi Oral
Number analyzed (Participants) | 6
Hours | 7.0000 [2.000 to 8.017]

7. Primary Outcome: Terminal Phase Half-life (t1/2) of Total Drug-related Material (Radioactivity) in Plasma for Treatment Period 1
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis.
Time Frame: as for outcome 1
Population: PK Population. Only those participants available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Nemi IH + 14C-Nemi IV
Number analyzed (Participants) | 3
Hours | 56.9152 (7.69827)

8. Primary Outcome: Terminal Phase Half-life (t1/2) of Total Drug-related Material (Radioactivity) in Plasma for Treatment Period 2
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis. NA indicates that data is not available as single participant was analyzed.
Time Frame: Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96 and 168 h post-dose
Population: PK Population. Only those participants available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | 14C-Nemi Oral
Number analyzed (Participants) | 1
Hours | 39.6279 (NA) — NA indicates that data is not available as single participant was analyzed

9. Primary Outcome: Urinary and Faecal Cumulative Excretion as a Percentage of the Total Radioactive Dose Administered Over Time for Treatment Period 1
Description: Urine samples and fecal samples were collected to measure total radiolabeled drug-related material excreted in urine and feces respectively.
Time Frame: Up to 168 hours
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Percentage of dose excreted
Arm/Group | Nemi IH + 14C-Nemi IV
Number analyzed (Participants) | 6
Percentage of dose excreted
  Fe Feces, 0 to 24 hour | 0.3961 (0.83271)
  Fe Feces, 24 to 48 hour | 2.1998 (3.77158)
  Fe Feces, 48 to 72 hour | 18.1265 (12.97670)
  Fe Feces, 72 to 96 hour | 28.0481 (18.22334)
  Fe Feces, 96 to 120 hour | 33.7465 (19.02044)
  Fe Feces, 120 to 144 hour | 45.2398 (14.63248)
  Fe Feces, 144 to 168 hour | 51.6981 (15.46780)
  Fe Urine, 0 to 6 hour | 2.1567 (0.83754)
  Fe Urine, 6 to 24 hour | 5.1183 (1.53825)
  Fe Urine, 24 to 48 hour | 7.6850 (2.04159)
  Fe Urine, 48 to 72 hour | 9.3483 (2.26387)
  Fe Urine, 72 to 96 hour | 10.7150 (2.46640)
  Fe Urine, 96 to 120 hour | 11.6400 (2.52790)
  Fe Urine, 120 to 144 hour | 12.3607 (2.56693)
  Fe Urine, 144 to 168 hour | 12.9205 (2.57056)
  Fe Total (Urine+Feces), 0 to 24 hour | 5.5145 (1.30554)
  Fe Total (Urine+Feces), 24 to 48 hour | 9.8848 (3.03062)
  Fe Total (Urine+Feces), 48 to 72 hour | 27.4748 (13.02973)
  Fe Total (Urine+Feces), 72 to 96 hour | 38.7631 (18.40877)
  Fe Total (Urine+Feces), 96 to 120 hour | 45.3865 (19.01459)
  Fe Total (Urine+Feces), 120 to 144 hour | 57.6005 (14.46954)
  Fe Total (Urine+Feces), 144 to 168 hour | 64.6186 (15.25339)

10. Primary Outcome: Urinary and Fecal Cumulative Excretion as a Percentage of the Total Radioactive Dose Administered Over Time for Treatment Period 2
Description: Urine samples and fecal samples were collected to measure total radiolabeled drug-related material excreted in urine and feces respectively. Only those participants available at the specified time points were analyzed represented by n=X in the category titles.
Time Frame: Up to 336 hours
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Percentage of dose excreted
Arm/Group | 14C-Nemi Oral
Number analyzed (Participants) | 6
Percentage of dose excreted
  Fe Feces, 0 to 24 hour; n=6 | 3.81330 (7.16484)
  Fe Feces, 24 to 48 hour; n=6 | 14.6367 (21.64607)
  Fe Feces, 48 to 72 hour; n=6 | 40.9583 (28.48392)
  Fe Feces, 72 to 96 hour; n=6 | 48.8217 (29.60581)
  Fe Feces, 96 to 120 hour; n=6 | 60.7617 (18.24192)
  Fe Feces, 120 to 144 hour; n=6 | 64.1667 (19.65337)
  Fe Feces, 144 to 168 hour; n=6 | 72.4217 (6.66365)
  Fe Feces, 168 to 192 hour; n=6 | 75.1117 (5.29605)
  Fe Feces, 192 to 216 hour; n=6 | 77.0917 (4.59090)
  Fe Feces, 216 to 240 hour; n=6 | 77.5933 (4.12513)
  Fe Feces, 240 to 264 hour; n=6 | 78.7917 (3.82906)
  Fe Feces, 264 to 288 hour; n=5: number analyzed (Participants) | 5
  Fe Feces, 264 to 288 hour; n=5 | 78.6820 (4.07492)
  Fe Feces, 288 to 312 hour; n=3: number analyzed (Participants) | 3
  Fe Feces, 288 to 312 hour; n=3 | 80.9500 (3.78747)
  Fe Feces, 312 to 336 hour; n=3: number analyzed (Participants) | 3
  Fe Feces, 312 to 336 hour; n=3 | 81.1500 (3.57979)
  Fe Urine, 0 to 6 hour; n=6 | 0.3867 (0.09668)
  Fe Urine, 6 to 24 hour; n=6 | 1.7017 (0.42995)
  Fe Urine, 24 to 48 hour; n=6 | 2.7183 (0.73249)
  Fe Urine, 48 to 72 hour; n=6 | 3.4250 (0.89063)
  Fe Urine, 72 to 96 hour; n=6 | 3.9600 (0.97980)
  Fe Urine, 96 to 120 hour; n=6 | 4.3617 (1.02918)
  Fe Urine, 120 to 144 hour; n=6 | 4.6717 (1.09549)
  Fe Urine, 144 to 168 hour; n=6 | 4.9217 (1.12583)
  Fe Urine, 168 to 192 hour; n=6 | 5.1383 (1.16426)
  Fe Urine, 192 to 216 hour; n=6 | 5.2950 (1.16156)
  Fe Urine, 216 to 240 hour; n=6 | 5.4700 (1.20854)
  Fe Urine, 240 to 264 hour; n=6 | 5.5617 (1.24856)
  Fe Urine, 264 to 288 hour; n=5: number analyzed (Participants) | 5
  Fe Urine, 264 to 288 hour; n=5 | 5.4760 (1.35858)
  Fe Urine, 288 to 312 hour; n=3: number analyzed (Participants) | 3
  Fe Urine, 288 to 312 hour; n=3 | 5.7800 (1.43293)
  Fe Urine, 312 to 336 hour; n=3: number analyzed (Participants) | 3
  Fe Urine, 312 to 336 hour; n=3 | 5.8133 (1.45590)
  Fe Total (Urine+Feces), 0 to 24 hour; n=6 | 5.5150 (7.01205)
  Fe Total (Urine+Feces), 24 to 48 hour; n=6 | 17.3550 (21.303)
  Fe Total (Urine+Feces), 48 to 72 hour; n=6 | 44.3833 (28.28365)
  Fe Total (Urine+Feces), 72 to 96 hour; n=6 | 52.7817 (29.36619)
  Fe Total (Urine+Feces), 96 to 120 hour; n=6 | 65.1233 (17.8525)
  Fe Total (Urine+Feces), 120 to 144 hour; n=6 | 68.8383 (19.24589)
  Fe Total (Urine+Feces), 144 to 168 hour; n=6 | 77.3433 (6.27302)
  Fe Total (Urine+Feces), 168 to 192 hour; n=6 | 80.2500 (4.74848)
  Fe Total (Urine+Feces), 192 to 216 hour; n=6 | 82.3867 (3.98209)
  Fe Total (Urine+Feces), 216 to 240 hour; n=6 | 83.0633 (3.3933)
  Fe Total (Urine+Feces), 240 to 264 hour; n=6 | 84.3533 (3.17528)
  Fe Total (Urine+Feces), 264 to 288 hour; n=5: number analyzed (Participants) | 5
  Fe Total (Urine+Feces), 264 to 288 hour; n=5 | 84.158 (3.25412)
  Fe Total (Urine+Feces), 288 to 312 hour; n=3: number analyzed (Participants) | 3
  Fe Total (Urine+Feces), 288 to 312 hour; n=3 | 86.7300 (2.44851)
  Fe Total (Urine+Feces), 312 to 336 hour; n=3: number analyzed (Participants) | 3
  Fe Total (Urine+Feces), 312 to 336 hour; n=3 | 86.9633 (2.16207)

11. Secondary Outcome: AUC (0 to Inf) and AUC (0 to t) of Parent GSK2269557 and [14C]-GSK2269557 in Plasma for Treatment Period 1
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis. For measured concentrations of GSK2269557 in blood plasma, the nomenclature [14C]-GSK2269557 describes the parent GSK2269557 concentration derived via analysis by LC+AMS, whereas GSK2269557 describes the parent GSK2269557 concentration derived via LC/MS. Only those participants available at the specified time points were analyzed represented by n=X in the category titles.
Time Frame: as for outcome 1
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*picogram per milliliter
Arm/Group | Nemi IH + 14C-Nemi IV
Number analyzed (Participants) | 6
Hour*picogram per milliliter
  GSK2269557: AUC (0 to inf), n=6 | 33374.56 (33.190)
  GSK2269557: AUC (0 to t), n=6 | 28425.82 (34.474)
  [14C]-GSK2269557: AUC (0 to inf), n=4: number analyzed (Participants) | 4
  [14C]-GSK2269557: AUC (0 to inf), n=4 | 750.5798 (48.27760)
  [14C]-GSK2269557: AUC (0 to t), n=6 | 546.4731 (45.31868)

12. Secondary Outcome: AUC (0 to Inf) and AUC (0 to t) of [14C]-GSK2269557 in Plasma for Treatment Period 2
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis. Only those participants with data available at the specified time points were analyzed represented by n=X in the category titles. For measured concentrations of GSK2269557 in blood plasma, the nomenclature [14C]-GSK2269557 describes the parent GSK2269557 concentration derived via analysis by LC+AMS.
Time Frame: Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96 and 168 h post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*picogram per milliliter
Arm/Group | 14C-Nemi Oral
Number analyzed (Participants) | 6
Hour*picogram per milliliter
  AUC (0 to inf), n=4: number analyzed (Participants) | 4
  AUC (0 to inf), n=4 | 25107.96 (46.310)
  AUC (0 to t), n=6 | 16913.06 (53.841)

13. Secondary Outcome: Cmax of Parent GSK2269557 and [14C]-GSK2269557 in Plasma for Treatment Period 1
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis. For measured concentrations of GSK2269557 in blood plasma, the nomenclature [14C]-GSK2269557 describes the parent GSK2269557 concentration derived via analysis by LC+AMS, whereas GSK2269557 describes the parent GSK2269557 concentration derived via LC/MS.
Time Frame: as for outcome 1
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picograms per milliliter
Arm/Group | Nemi IH + 14C-Nemi IV
Number analyzed (Participants) | 6
Picograms per milliliter
  GSK2269557 | 5258.98 (62.819)
  [14C]-GSK2269557 | 205.6264 (57.91419)

14. Secondary Outcome: Cmax of [14C]-GSK2269557 in Plasma for Treatment Period 2
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis. For measured concentrations of GSK2269557 in blood plasma, the nomenclature [14C]-GSK2269557 describes the parent GSK2269557 concentration derived via analysis by LC+AMS.
Time Frame: Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96 and 168 h post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picograms per milliliter
Arm/Group | 14C-Nemi Oral
Number analyzed (Participants) | 6
Picograms per milliliter | 398.8822 (27.81929)

15. Secondary Outcome: Tmax of Parent GSK2269557 and [14C]-GSK2269557 in Plasma for Treatment Period 1
Description: as for outcome 13
Time Frame: as for outcome 1
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Nemi IH + 14C-Nemi IV
Number analyzed (Participants) | 6
Hours
  GSK2269557 | 0.0333 [0.017 to 0.050]
  [14C]-GSK2269557 | 0.2333 [0.2333 to 0.2333]

16. Secondary Outcome: Tmax of [14C]-GSK2269557 in Plasma for Treatment Period 2
Description: as for outcome 14
Time Frame: Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96 and 168 h post-dose
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | 14C-Nemi Oral
Number analyzed (Participants) | 6
Hours | 6.0000 [2.000 to 8.000]

17. Secondary Outcome: t1/2 of Parent GSK2269557 and [14C]-GSK2269557 in Plasma for Treatment Period 1
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis. For measured concentrations of GSK2269557 in blood plasma, the nomenclature [14C]-GSK2269557 describes the parent GSK2269557 concentration derived via analysis by LC+AMS, whereas GSK2269557 describes the parent GSK2269557 concentration derived via LC/MS. Only those participants available at the indicated time points were analyzed represented by n=X in the category titles.
Time Frame: as for outcome 1
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Nemi IH + 14C-Nemi IV
Number analyzed (Participants) | 6
Hours
  GSK2269557 | 58.4408 (16.84150)
  [14C]-GSK2269557 | 54.7223 (35.98970)

18. Secondary Outcome: t1/2 of [14C]-GSK2269557 in Plasma for Treatment Period 2
Description: as for outcome 14
Time Frame: Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96 and 168 h post-dose
Population: PK Population. Only those participants available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | 14C-Nemi Oral
Number analyzed (Participants) | 4
Hours | 50.8028 (40.16665)

19. Secondary Outcome: Volume of Distribution of Parent [14C]-GSK2269557 After IV Dose Only in Plasma
Description: as for outcome 14
Time Frame: as for outcome 1
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Nemi IH + 14C-Nemi IV
Number analyzed (Participants) | 4
Liters
  Vss | 727.7102 (11.24581)
  Vz | 851.4423 (13.98220)

20. Secondary Outcome: Clearance of Parent [14C]-GSK2269557 After IV Dose Only in Plasma
Description: as for outcome 14
Time Frame: as for outcome 1
Population: PK Population. Only those participants available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Nemi IH + 14C-Nemi IV
Number analyzed (Participants) | 4
Liters per hour | 10.7849 (46.70161)

21. Secondary Outcome: Inhaled Absolute Bioavailability (F) for Treatment Period 1
Description: Absolute bioavailability (F) was estimated for the inhaled doses for each participant and is reported. Only those participants available at the specified time points were analyzed represented by n=X in the category titles.
Time Frame: as for outcome 1
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Fraction of drug
Arm/Group | Nemi IH + 14C-Nemi IV
Number analyzed (Participants) | 6
Fraction of drug
  Inhaled F (0 to inf); n=4: number analyzed (Participants) | 4
  Inhaled F (0 to inf); n=4 | 0.3807 (19.65374)
  Inhaled F (0 to t); n=6 | 0.4213 (21.84410)

22. Secondary Outcome: Oral Absolute Bioavailability (F) for Treatment Period 2
Description: Absolute bioavailability (F) was estimated for the oral doses for each participant and is reported. Only those participants available at the specified time points were analyzed represented by n=X in the category titles.
Time Frame: Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96 and 168 h post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Fraction of drug
Arm/Group | 14C-Nemi Oral
Number analyzed (Participants) | 6
Fraction of drug
  Oral F (0 to inf); n=4: number analyzed (Participants) | 4
  Oral F (0 to inf); n=4 | 0.3515 (3.35095)
  Oral F (0 to t); n=6 | 0.3261 (12.77892)

23. Secondary Outcome: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with use of a medicinal product (MP), whether or not considered related to MP. AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with use of MP. SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant or all events of possible drug induced liver injury with hyperbilirubinemia.
Time Frame: Up to 11 weeks
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Groups:
- 14C-Nemi Oral: Participants received solution of [14C] radiolabelled GSK2269557 as a single dose of 800 µg, administered as an oral solution.
Arm/Group | Nemi IH + 14C-Nemi IV | 14C-Nemi Oral
Number analyzed (Participants) | 6 | 6
Participants
  AE | 0 | 1
  SAE | 0 | 0

24. Secondary Outcome: Number of Participants With Hematology Parameters of Potential Clinical Concern
Description: Hematology parameters included basophils, eosinophils, erythrocytes, monocytes, hematocrit, hemoglobin, lymphocytes, neutrophil count, platelet count and white blood cells. Number of participants with hematology parameters of potential clinical concern are presented.
Time Frame: Up to 11 weeks
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Nemi IH + 14C-Nemi IV | 14C-Nemi Oral
Number analyzed (Participants) | 6 | 6
Participants | 2 | 1

25. Secondary Outcome: Number of Participants With Clinical Chemistry Parameters of Potential Clinical Concern
Description: Clinical chemistry parameters included alanine aminotransferase, alkaline phosphatase, aspartate aminotransferase, bilirubin, chloride, cholesterol, gamma glutamyl transferase, globulin, protein, triglycerides, urate, albumin, calcium, creatinine, glucose, phosphorous, potassium, urea and sodium. Number of participants with clinical chemistry parameters of potential clinical concern are presented.
Time Frame: Up to 11 weeks
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Nemi IH + 14C-Nemi IV | 14C-Nemi Oral
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

26. Secondary Outcome: Number of Participants With Clinically Significant Urinalysis Findings
Description: Urine samples were collected to detect the presence of bilirubin, glucose, ketones, leukocyte esterase, nitrite, occult blood, protein and urobilinogen. Urinalysis also included measurement of specific gravity and pH. Number of participants with clinically significant urinalysis findings are presented.
Time Frame: Up to 168 hours
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Nemi IH + 14C-Nemi IV | 14C-Nemi Oral
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

27. Secondary Outcome: Number of Participants With Electrocardiogram Findings of Clinical Significance
Description: Twelve-lead electrocardiogram was measured in a supine or semi-supine position after 5 minutes rest. Number of participants with electrocardiogram findings of clinical significance are presented.
Time Frame: Up to 11 weeks
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Nemi IH + 14C-Nemi IV | 14C-Nemi Oral
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

28. Secondary Outcome: Number of Participants With Vital Signs of Potential Clinical Concern
Description: Vital signs were measured in a supine or semi-supine position after 5 minutes rest and included temperature, systolic and diastolic blood pressure and pulse and respiratory rate. Number of participants with vital signs of potential clinical concern are reported.
Time Frame: Up to 11 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Nemi IH + 14C-Nemi IV | 14C-Nemi Oral
Number analyzed (Participants) | 6 | 6
Participants
  High respiratory rate | 1 | 0
  Low temperature | 1 | 0

ADVERSE EVENTS:
Time Frame: Serious and non serious adverse events were evaluated up to 11 weeks
Description: Safety Population was analyzed to collect serious adverse events (SAE) and non-serious adverse events (nSAE).
Groups:
- 14C-Nemi Oral: Participants received solution of [14C] radiolabelled GSK2269557 as a single dose of 800 µg orally
Arm/Group | Nemi IH + 14C-Nemi IV | 14C-Nemi Oral
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nemi IH + 14C-Nemi IV (N=6) | 14C-Nemi Oral (N=6)
Malaise (General disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-10-30): https://cdn.clinicaltrials.gov/large-docs/59/NCT03315559/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-09): https://cdn.clinicaltrials.gov/large-docs/59/NCT03315559/SAP_001.pdf